CLINICAL TRIAL: NCT00992511
Title: Immunological Non-inferiority Between Two Process-manufactured Influenza Vaccines in Adults Aged 18 to 60 Years
Brief Title: Study to Evaluate the Immunogenicity and Safety of an Investigational Influenza (H1N1 Influenza Virus) Vaccine in Adults, Using Two Different Manufacturing Processes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113809
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- GSK2340272A New 1D Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received one dose of the New process-manufactured (New 1D) GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
  Interventions: Biological: GSK investigational vaccine GSK2340272A
- GSK2340272A New 2D Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of the New process-manufactured (New 2D) GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: GSK investigational vaccine GSK2340272A
- GSK2340272A INI 1D Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received one dose of the Initial process-manufactured (INI 1D) GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
  Interventions: Biological: GSK investigational vaccine GSK2340272A
- GSK2340272A INI 2D Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of the Initial process-manufactured (INI 2D) GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: GSK investigational vaccine GSK2340272A

INTERVENTIONS:
Biological: GSK investigational vaccine GSK2340272A — One intramuscular injection of initial process-manufactured GSK2340272A vaccine
  Arms: GSK2340272A New 1D Group
Biological: GSK investigational vaccine GSK2340272A — Two intramuscular injections of initial process-manufactured GSK2340272A vaccine
  Arms: GSK2340272A New 2D Group
Biological: GSK investigational vaccine GSK2340272A — One intramuscular injection of new process-manufactured GSK2340272A vaccine
  Arms: GSK2340272A INI 1D Group
Biological: GSK investigational vaccine GSK2340272A — Two intramuscular injections of new process-manufactured GSK2340272A vaccine
  Arms: GSK2340272A INI 2D Group

SUMMARY:
The objective of this study is to evaluate the immunogenicity and safety of one or two doses of GSK Biologicals' investigational influenza vaccine GSK2340272A, manufactured using two different processes, in adults aged 18 to 60 years.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must satisfy ALL the following criteria at study entry:
* A male or female aged 18 to 60 years of age at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study. Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5°C (99.5°F), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with coumarin derivatives, other vitamin K antagonists or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* Any contraindication to intramuscular administration of the influenza vaccines.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-10-14 (Actual); Primary Completion 2010-11-09 (Actual); Study Completion 2010-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (3):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113809 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Started | 76 | 73 | 76 | 75
Completed | 74 | 73 | 74 | 70
Not Completed | 2 | 0 | 2 | 5
Not completed — Migrated/moved from study area | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group | Total
Number analyzed (Participants) | 76 | 73 | 76 | 75 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (13.02) | 40.9 (12.20) | 40.5 (12.45) | 38.6 (12.10) | 39.84 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 43 | 38 | 162
  Male | 34 | 34 | 33 | 37 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic/North African heritage | 0 | 0 | 0 | 1 | 1
  White - Caucasian/European heritage | 76 | 73 | 76 | 74 | 299

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Were Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:10, that usually is accepted as indicating protection.
Time Frame: At Day 21
Population: The According-to Protocol (ATP) cohort for immunogenicity included all evaluable subjects for whom one or two doses were taken and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after each vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 74 | 64 | 69 | 63
Participants | 74 | 64 | 69 | 63

2. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 74 | 64 | 69 | 63
Titers | 323.0 [253.4 to 411.8] | 334.2 [267.9 to 416.9] | 341.5 [261.7 to 445.6] | 398.9 [294.8 to 539.7]
Statistical Analysis 1: Comparison: GSK2340272A New 1D Group vs GSK2340272A INI 1D Group; To evaluate the immunological non-inferiority (in terms of vaccine-homologous virus H1N1 Haemagglutinin Inhibition [HI] antibody geometric mean titres [GMTs]) of the new process-manufactured A/California/7/2009 (H1N1)v-like antigen compared to the initial process-manufactured A/California/7/2009 (H1N1)v-like antigen, 21 days after first vaccination in healthy subjects aged 18 to 60 years; Test type: Non-Inferiority — Criterion for non-inferiority: upper limit (UL) of the two-sided 95% Confidence Interval (CI) for the ratio of GMT between the initial process-manufactured vaccine (GSK2340272A INI 2D Group) and (over) new process-manufactured vaccine (GSK2340272A NEW 2D Group) was less than or equal to (≤) 2; Adjusted GMT ratio = 1.06, 95% CI 2-sided [0.77 to 1.46]
Statistical Analysis 2: Comparison: GSK2340272A New 2D Group vs GSK2340272A INI 2D Group; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Adjusted GMT ratio = 1.17, 95% CI 2-sided [0.86 to 1.61]

3. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection.
Time Frame: At Days 0 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 74 | 64 | 71 | 63
Participants
  Flu A/CAL/7/09, Day 0 | 28 | 23 | 30 | 22
  Flu A/CAL/7/09, Day 42 | 74 | 64 | 71 | 62

4. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 2
Time Frame: At Days 0 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 74 | 64 | 71 | 63
Titer
  Flu A/CAL/7/09, Day 0 | 8.6 [7.0 to 10.6] | 8.0 [6.7 to 9.6] | 8.9 [7.2 to 11.0] | 8.4 [6.8 to 10.3]
  Flu A/CAL/7/09, Day 42 | 226.4 [176.8 to 289.8] | 470.0 [387.9 to 569.6] | 268.4 [206.2 to 349.3] | 676.8 [564.7 to 811.3]

5. Secondary Outcome: Number of Subjects Who Were Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 1
Time Frame: At Days 182 and 364
Population: The ATP cohort for antibody persistence at Day 182 and 364 included all evaluable subjects for whom one or two doses were taken and for whom data concerning immunogenicity outcome measures were available. This cohort included subjects for whom assay results were available for antibodies against the study vaccine antigen component at Day 182 and 364
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 72 | 68 | 69 | 65
Participants
  Flu A/California/7/2009, Day 182 | 71 | 68 | 68 | 65
  Flu A/California/7/2009, Day 364: number analyzed (Participants) | 65 | 63 | 62 | 58
  Flu A/California/7/2009, Day 364 | 64 | 63 | 60 | 58

6. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: as for outcome 2
Time Frame: At Days 182 and 364
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 72 | 68 | 69 | 65
Titers
  Flu A/California/7/2009, Day 182 | 102.7 [79.4 to 132.9] | 147.5 [120.9 to 180.0] | 128.3 [94.9 to 173.3] | 226.3 [183.5 to 279.1]
  Flu A/California/7/2009, Day 364: number analyzed (Participants) | 65 | 63 | 62 | 58
  Flu A/California/7/2009, Day 364 | 63.9 [48.8 to 83.7] | 75.7 [59.8 to 96.0] | 81.3 [58.6 to 112.7] | 123.7 [95.2 to 160.8]

7. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 post vaccination], antibody titer greater than or equal to (≥) 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 74 | 64 | 71 | 63
Participants
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 74 | 64 | 69 | 63
  Flu A/CAL/7/09, Day 21 | 71 | 62 | 65 | 61
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 74 | 64 | 71 | 62
  Flu A/CAL/7/09, Day 42 | 68 | 62 | 65 | 62

8. Secondary Outcome: Number of SCR Subjects for HI Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 post to vaccination], antibody titer greater than or equal to (≥) 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Days 182 and 364
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 72 | 68 | 69 | 65
Participants
  Flu A/CAL/7/09, Day 182 | 60 | 63 | 55 | 64
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 65 | 63 | 62 | 58
  Flu A/CAL/7/09, Day 364 | 43 | 49 | 41 | 50

9. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 3
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 74 | 64 | 71 | 63
Participants
  Flu A/CAL/7/09, Day 0 | 6 | 4 | 6 | 2
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 74 | 64 | 69 | 63
  Flu A/CAL/7/09, Day 21 | 73 | 64 | 67 | 62
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 74 | 64 | 71 | 62
  Flu A/CAL/7/09, Day 42 | 71 | 64 | 68 | 62

10. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 3
Time Frame: At Days 182 and 364
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 72 | 68 | 69 | 65
Participants
  Flu A/CAL/7/09, Day 182 | 63 | 66 | 60 | 65
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 65 | 63 | 62 | 58
  Flu A/CAL/7/09, Day 364 | 47 | 54 | 48 | 53

11. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 74 | 64 | 71 | 63
Fold increase
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 74 | 64 | 69 | 63
  Flu A/CAL/7/09, Day 21 | 37.4 [28.8 to 48.6] | 41.8 [31.5 to 55.3] | 38.0 [28.3 to 51.0] | 47.7 [35.7 to 63.7]
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 74 | 64 | 71 | 62
  Flu A/CAL/7/09, Day 42 | 26.2 [20.2 to 33.9] | 58.7 [44.6 to 77.3] | 30.1 [22.6 to 40.0] | 82.5 [66.4 to 102.5]

12. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 11
Time Frame: At Days 182 and 364
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 72 | 68 | 69 | 65
Fold increase
  Flu A/CAL/7/09, Day 182 | 12.1 [9.6 to 15.3] | 18.9 [15.3 to 23.5] | 14.3 [10.6 to 19.2] | 25.6 [20.9 to 31.5]
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 65 | 63 | 62 | 58
  Flu A/CAL/7/09, Day 364 | 7.6 [6.0 to 9.8] | 9.5 [7.6 to 11.9] | 8.9 [6.4 to 12.5] | 13.5 [10.7 to 17.0]

13. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest; prevented normal activities as assessed by inability to attend/do work or school. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 76 | 73 | 74 | 75
Participants
  Any Pain, Dose 1 | 71 | 62 | 69 | 66
  Grade 3 Pain, Dose 1 | 2 | 2 | 1 | 2
  Any Redness, Dose 1 | 1 | 1 | 4 | 1
  Grade 3 Redness, Dose 1 | 1 | 0 | 0 | 0
  Any Swelling, Dose 1 | 4 | 4 | 3 | 7
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Pain, Dose 2 | 0 | 61 | 0 | 59
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Pain, Dose 2 | 0 | 0 | 0 | 3
  Any Redness, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Redness, Dose 2 | 0 | 3 | 0 | 3
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Swelling, Dose 2 | 0 | 5 | 0 | 7
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 71 | 67 | 69 | 68
  Grade 3 Pain, Across doses | 2 | 2 | 1 | 5
  Any Redness, Across doses | 1 | 3 | 4 | 4
  Grade 3 Redness, Across doses | 1 | 0 | 0 | 0
  Any Swelling, Across doses | 4 | 7 | 3 | 11
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and overall
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 71 | 67 | 69 | 68
Days
  Pain, Dose 1: number analyzed (Participants) | 71 | 62 | 69 | 66
  Pain, Dose 1 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 4.0]
  Pain, Dose 2: number analyzed (Participants) | 0 | 61 | 0 | 59
  Pain, Dose 2 |  | 3.0 [2.0 to 3.0] |  | 3.0 [2.0 to 3.0]
  Pain, Overall/dose | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 4.0]
  Redness, Dose 1: number analyzed (Participants) | 1 | 1 | 4 | 1
  Redness, Dose 1 | 5.0 [5.0 to 5.0] | 2.0 [2.0 to 2.0] | 1.5 [1.0 to 3.0] | 2.0 [2.0 to 2.0]
  Redness, Dose 2: number analyzed (Participants) | 0 | 3 | 0 | 3
  Redness, Dose 2 |  | 2.0 [1.0 to 5.0] |  | 4.0 [2.0 to 5.0]
  Redness, Overall/dose: number analyzed (Participants) | 1 | 3 | 4 | 4
  Redness, Overall/dose | 5.0 [5.0 to 5.0] | 2.0 [1.5 to 3.5] | 1.5 [1.0 to 3.0] | 3.0 [2.0 to 4.5]
  Swelling, Dose 1: number analyzed (Participants) | 4 | 4 | 3 | 7
  Swelling, Dose 1 | 4.0 [3.0 to 5.0] | 3.0 [2.0 to 3.5] | 1.0 [1.0 to 5.0] | 3.0 [2.0 to 5.0]
  Swelling, Dose 2: number analyzed (Participants) | 0 | 5 | 0 | 7
  Swelling, Dose 2 |  | 3.0 [2.0 to 3.0] |  | 2.0 [2.0 to 4.0]
  Swelling, Overall/dose: number analyzed (Participants) | 4 | 7 | 3 | 11
  Swelling, Overall/dose | 4.0 [3.0 to 5.0] | 3.0 [2.0 to 3.0] | 1.0 [1.0 to 5.0] | 2.5 [2.0 to 4.0]

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = temperature > 39.0 °C and ≤ 40°C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 76 | 73 | 74 | 75
Participants
  Any Fatigue, Dose 1 | 19 | 30 | 19 | 31
  Grade 3 Fatigue, Dose 1 | 1 | 2 | 0 | 2
  Related Fatigue, Dose 1 | 17 | 22 | 17 | 29
  Any Headache, Dose 1 | 25 | 22 | 21 | 31
  Grade 3 Headache, Dose 1 | 0 | 2 | 0 | 3
  Related Headache, Dose 1 | 18 | 17 | 15 | 27
  Any Joint pain, Dose 1 | 13 | 14 | 9 | 15
  Grade 3 Joint pain, Dose 1 | 1 | 1 | 0 | 1
  Related Joint pain, Dose 1 | 13 | 12 | 6 | 14
  Any Muscle aches, Dose 1 | 26 | 22 | 25 | 28
  Grade 3 Muscle aches, Dose 1 | 1 | 1 | 1 | 0
  Related Muscle aches, Dose 1 | 24 | 20 | 17 | 28
  Any Shivering, Dose 1 | 9 | 19 | 12 | 29
  Grade 3 Shivering, Dose 1 | 0 | 0 | 1 | 2
  Related Shivering, Dose 1 | 8 | 16 | 10 | 27
  Any Sweating, Dose 1 | 7 | 9 | 6 | 12
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 2
  Related Sweating, Dose 1 | 5 | 4 | 5 | 10
  Any Temperature, Dose 1 | 2 | 1 | 2 | 2
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0
  Related Temperature, Dose 1 | 2 | 1 | 2 | 2
  Any Fatigue, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Fatigue, Dose 2 | 0 | 29 | 0 | 33
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Fatigue, Dose 2 | 0 | 2 | 0 | 2
  Related Fatigue, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Related Fatigue, Dose 2 | 0 | 27 | 0 | 26
  Any Headache, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Headache, Dose 2 | 0 | 24 | 0 | 32
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Headache, Dose 2 | 0 | 2 | 0 | 3
  Related Headache, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Related Headache, Dose 2 | 0 | 17 | 0 | 26
  Any Joint pain, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Joint pain, Dose 2 | 0 | 15 | 0 | 22
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Joint pain, Dose 2 | 0 | 1 | 0 | 3
  Related Joint pain, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Related Joint pain, Dose 2 | 0 | 15 | 0 | 19
  Any Muscle aches, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Muscle aches, Dose 2 | 0 | 21 | 0 | 26
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Muscle aches, Dose 2 | 0 | 1 | 0 | 3
  Related Muscle aches, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Related Muscle aches, Dose 2 | 0 | 21 | 0 | 26
  Any Shivering, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Shivering, Dose 2 | 0 | 21 | 0 | 21
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Shivering, Dose 2 | 0 | 2 | 0 | 4
  Related Shivering, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Related Shivering, Dose 2 | 0 | 21 | 0 | 18
  Any Sweating, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Sweating, Dose 2 | 0 | 10 | 0 | 10
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Sweating, Dose 2 | 0 | 1 | 0 | 1
  Related Sweating, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Related Sweating, Dose 2 | 0 | 9 | 0 | 9
  Any Temperature, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Any Temperature, Dose 2 | 0 | 4 | 0 | 5
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Grade 3 Temperature, Dose 2 | 0 | 1 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 0 | 70 | 0 | 71
  Related Temperature, Dose 2 | 0 | 4 | 0 | 5
  Any Fatigue, Across doses | 19 | 43 | 19 | 43
  Grade 3 Fatigue, Across doses | 1 | 4 | 0 | 4
  Related Fatigue, Across doses | 17 | 36 | 17 | 38
  Any Headache, Across doses | 25 | 36 | 21 | 43
  Grade 3 Headache, Across doses | 0 | 4 | 0 | 5
  Related Headache, Across doses | 18 | 26 | 15 | 36
  Any Joint pain, Across doses | 13 | 23 | 9 | 27
  Grade 3 Joint pain, Across doses | 1 | 2 | 0 | 4
  Related Joint pain, Across doses | 13 | 22 | 6 | 23
  Any Muscle aches, Across doses | 26 | 35 | 25 | 37
  Grade 3 Muscle aches, Across doses | 1 | 2 | 1 | 3
  Related Muscle aches, Across doses | 24 | 33 | 17 | 37
  Any Shivering, Across doses | 9 | 33 | 12 | 40
  Grade 3 Shivering, Across doses | 0 | 2 | 1 | 6
  Related Shivering, Across doses | 8 | 30 | 10 | 35
  Any Sweating, Across doses | 7 | 17 | 6 | 20
  Grade 3 Sweating, Across doses | 0 | 1 | 0 | 3
  Related Sweating, Across doses | 5 | 13 | 5 | 17
  Any Temperature, Across doses | 2 | 5 | 2 | 6
  Grade 3 Temperature, Across doses | 0 | 1 | 0 | 0
  Related Temperature, Across doses | 2 | 5 | 2 | 6

16. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and overall
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 76 | 73 | 74 | 75
Days
  Fatigue, Dose 1: number analyzed (Participants) | 19 | 30 | 19 | 31
  Fatigue, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Fatigue, Dose 2: number analyzed (Participants) | 0 | 29 | 0 | 33
  Fatigue, Dose 2 |  | 2.0 [1.0 to 2.0] |  | 2.0 [1.0 to 3.0]
  Fatigue, Overall/dose: number analyzed (Participants) | 19 | 43 | 19 | 43
  Fatigue, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Headache, Dose 1: number analyzed (Participants) | 25 | 22 | 21 | 31
  Headache, Dose 1 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache, Dose 2: number analyzed (Participants) | 0 | 24 | 0 | 32
  Headache, Dose 2 |  | 1.0 [1.0 to 2.0] |  | 2.0 [1.0 to 3.0]
  Headache, Overall/dose: number analyzed (Participants) | 25 | 36 | 21 | 43
  Headache, Overall/dose | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Joint pain, Dose 1: number analyzed (Participants) | 13 | 14 | 9 | 15
  Joint pain, Dose 1 | 2.0 [1.0 to 2.0] | 2.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Joint pain, Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 22
  Joint pain, Dose 2 |  | 2.0 [1.0 to 3.0] |  | 1.0 [1.0 to 2.0]
  Joint pain, Overall/dose: number analyzed (Participants) | 13 | 23 | 9 | 27
  Joint pain, Overall/dose | 2.0 [1.0 to 2.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Muscle aches, Dose 1: number analyzed (Participants) | 26 | 22 | 25 | 28
  Muscle aches, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0]
  Muscle aches, Dose 2: number analyzed (Participants) | 0 | 21 | 0 | 26
  Muscle aches, Dose 2 |  | 2.0 [1.0 to 3.0] |  | 3.0 [1.0 to 3.0]
  Muscle aches, Overall/dose: number analyzed (Participants) | 26 | 35 | 25 | 37
  Muscle aches, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0]
  Sweating, Dose 1: number analyzed (Participants) | 7 | 9 | 6 | 12
  Sweating, Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 4.0 [2.0 to 5.0] | 2.0 [1.0 to 2.5]
  Sweating, Dose 2: number analyzed (Participants) | 0 | 10 | 0 | 10
  Sweating, Dose 2 |  | 1.0 [1.0 to 2.0] |  | 1.0 [1.0 to 1.0]
  Sweating, Overall/dose: number analyzed (Participants) | 7 | 17 | 6 | 20
  Sweating, Overall/dose | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 4.0 [2.0 to 5.0] | 1.0 [1.0 to 2.0]
  Shivering, Dose 1: number analyzed (Participants) | 9 | 19 | 12 | 29
  Shivering, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering, Dose 2: number analyzed (Participants) | 0 | 21 | 0 | 21
  Shivering, Dose 2 |  | 1.0 [1.0 to 2.0] |  | 1.0 [1.0 to 2.0]
  Shivering, Overall/dose: number analyzed (Participants) | 9 | 33 | 12 | 40
  Shivering, Overall/dose | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Temperature, Dose 1: number analyzed (Participants) | 2 | 1 | 2 | 2
  Temperature, Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Temperature, Dose 2: number analyzed (Participants) | 0 | 4 | 0 | 5
  Temperature, Dose 2 |  | 1.5 [1.0 to 2.5] |  | 1.0 [1.0 to 1.0]
  Temperature, Overall/dose: number analyzed (Participants) | 2 | 5 | 2 | 6
  Temperature, Overall/dose | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

17. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: Any pIMD was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration. Related pIMD was defined as an event assessed by the investigator as possibly related to the study vaccination.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 76 | 73 | 76 | 75
Participants
  Any | 0 | 0 | 0 | 0
  Related | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 21 days after the first vaccination and 63 days after the second vaccination (Day 0 - Day 20 and Day 21 - Day 84)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 76 | 73 | 76 | 75
Participants
  Any AE(s), Days 0-20 | 17 | 20 | 28 | 18
  Grade 3 AE(s), Days 0-20 | 2 | 2 | 2 | 1
  Related AE(s), Days 0-20 | 5 | 13 | 5 | 4
  Any AE(s), up to Day 84: number analyzed (Participants) | 0 | 73 | 0 | 75
  Any AE(s), up to Day 84 | 0 | 30 | 0 | 35
  Grade 3 AE(s), up to Day 84: number analyzed (Participants) | 0 | 73 | 0 | 75
  Grade 3 AE(s), up to Day 84 | 0 | 7 | 0 | 6
  Related AE(s), up to Day 84: number analyzed (Participants) | 0 | 73 | 0 | 75
  Related AE(s), up to Day 84 | 0 | 15 | 0 | 7

19. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
Number analyzed (Participants) | 76 | 73 | 76 | 75
Participants | 7 | 2 | 3 | 5

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 84-day (Days 0-83) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 364).
Arm/Group | GSK2340272A New 1D Group | GSK2340272A New 2D Group | GSK2340272A INI 1D Group | GSK2340272A INI 2D Group
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/73 | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 7/76 | 2/73 | 3/76 | 5/75
Other Adverse Events (participants affected / at risk) | 72/76 | 70/73 | 71/76 | 71/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A New 1D Group (N=76) | GSK2340272A New 2D Group (N=73) | GSK2340272A INI 1D Group (N=76) | GSK2340272A INI 2D Group (N=75)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salpingitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A New 1D Group (N=76) | GSK2340272A New 2D Group (N=73) | GSK2340272A INI 1D Group (N=76) | GSK2340272A INI 2D Group (N=75)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 23 (31) | 9 (9) | 28 (39)
Chills (General disorders) | 9 (9) | 33 (40) | 12 (12) | 40 (50)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 4 (4) | 4 (4)
Fatigue (General disorders) | 19 (19) | 43 (61) | 19 (19) | 43 (65)
Headache (Nervous system disorders) | 25 (26) | 38 (56) | 23 (27) | 45 (77)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 17 (19) | 6 (6) | 20 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 26 (26) | 35 (43) | 25 (25) | 38 (55)
Nasopharyngitis (Infections and infestations) | 19 (19) | 7 (7) | 8 (8) | 11 (11)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 71 (71) | 67 (123) | 69 (69) | 68 (125)
Pyrexia (General disorders) | 3 (3) | 9 (10) | 3 (3) | 15 (17)
Swelling (General disorders) | 4 (4) | 7 (9) | 3 (3) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.